CLINICAL TRIAL: NCT00337805
Title: A Randomized Trial of Synthetic vs Normal Saline for the Flow-based Algorithmic Hemodynamic Resuscitation of Patients Post-cardiac Surgery
Brief Title: Double Blind Randomized Trial of Saline vs Pentaspan for Resuscitation After Cardiac Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Dr S Magder, McGill University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BMA-04-016
Record Dates: First submitted 2006-06-14; First posted 2006-06-16 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Cardiac Surgery
Keywords: colloid; crystalloid; hemodynamics; flow-directed; resuscitation
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 colloid (Active Comparator): Boluses of fluids are a pentastarch (up to 1000 ml)
  Interventions: Other: Pentaspan
- 2. Crytalloid (Active Comparator): Boluses are given as normal saline
  Interventions: Other: Pentaspan

INTERVENTIONS:
Other: Pentaspan — When fluids are indicated either pentaspan or saline are given in a double blind randomized assignment

SUMMARY:
This is a randomized double blind trial of the use of the use of colloids vs crystalloid solutions for resuscitation of patients after cardiac surgery. Patients are managed with an algorithm driven protocol that is based on the flow response to fluid challenges. The hypothesis is that the use of a colloid solution will result in less use of catecholamines at 8:00 the morning following surgery. Secondary end-points include total use of catecholamines, time in the ICU, return to the ICU, and safety issues including bleeding and renal function.

ELIGIBILITY:
Inclusion Criteria:

* status post cardiac surgery
* pulmonary artery occlusion catheter in place
* informed consent
* morning case (must be out of OR by 2:00 PM

Exclusion Criteria:

* excessive bleeding (> 200 cc/hr)
* intraaortic balloon pump
* refusal by treating team
* emergency cases
* patients with known adverse reactions to starch solutions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2004-09; Primary Completion 2007-12 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Use of catecholamines at 8:00 the morning after surgery | first post operative day

SECONDARY OUTCOMES:
Total use of catecholamines | Time in ICU
Time in the ICU | Time in ICU
Post-operative complications | Hospital stay or 28 days
Bleeding | Hospital stay or 28 days
Renal failure | Hospital stay or 28 days

CONTACTS AND LOCATIONS:
Overall Officials: sheldon magder, md, Principal Investigator — McGill University
Locations (1):
- Royal Victoria Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Potter BJ, Deverenne B, Doucette S, Fergusson D, Magder S; Canadian Critical Care Trials Group. Cardiac output responses in a flow-driven protocol of resuscitation following cardiac surgery. J Crit Care. 2013 Jun;28(3):265-9. doi: 10.1016/j.jcrc.2012.09.008. Epub 2012 Nov 14. PMID 23159133